CLINICAL TRIAL: NCT02850380
Title: Spatial Orientation and Motor Skills: How to Flip Switches "Down" in Weightlessness?
Acronym: Down
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: Novespace (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2015-A01261-48
Record Dates: First submitted 2016-04-21; First posted 2016-08-01 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Weightlessness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- spatial orientation in weightlessness (Other): subjects will be asked to flip a series of switches into the "off" position. On Earth, the "off" position corresponds to "down" in all three reference frames: the visual allocentric, the non-visual allocentric as well as the egocentric frames. We expect that flip direction will be dominated by visual allocentric cues when those are available, will be delayed and more variable when confirmatory gravitational cues are absent, and will be biased towards the egocentric reference when tactile cues are added
  Interventions: Other: FLIP SWITCHES "DOWN" IN WEIGHTLESSNESS

INTERVENTIONS:
Other: FLIP SWITCHES "DOWN" IN WEIGHTLESSNESS — The circular instrument panel that subjects will see into the cylindrical mask consists of one switch surrounded by a luminous ring (left part of the figure below). The switch can be flipped into any direction within the full 360° range. The switch provides no visual cues about "down", but the experimenter can add such cues by means of visually polarized labelling displayed on a circular black screen at the center of the panel (right part the figure below).

SUMMARY:
The purpose of the study is to investigate spatial orientation in weightlessness as it manifests not in perception but rather in motor performance by direction and reaction time of flip switch.

Hypotheses are that flip switch:

1. will be biased towards visual allocentric cues when those are available;
2. will be biased towards the egocentric reference when tactile cues are added;
3. will be dominated by egocentric cues when visual cues are not available;
4. will be delayed and more variable when confirmatory gravitational cues are absent;
5. will be faster and more reliable in absence of conflicting gravitational cues, and even more so when tactile cues are added;
6. The difference will be more pronounce when tested under Dual-task condition

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (men or women)
* Aged from 20 to 65
* Affiliated to a Social Security system and, for non-French resident, holding a European Health Insurance Card (EHIC)
* Who accepted to take part in the study
* Who have given their written stated consent
* Who has passed a medical examination similar to a standard aviation medical examination for private pilot aptitude (JAR FCL3 Class 2 medical examination). There will be no additional test performed for subject selection.

Subjects will be staff member of the team or of other teams participating in the parabolic flight campaign

Exclusion Criteria:

* Person who took part in a previous biomedical research protocol, of which exclusion period is not terminated
* Person who has already participated in a parabolic flight
* Pregnant women

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
reaction time of flip switch measured with a chronometer | baseline
Direction of flip switch measured with the circular instrument panel | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Pierre DP Denise, PhD, Principal Investigator — CHU CAEN
Locations (1):
- Caen CHU, Caen, France

IPD SHARING:
Plan to Share IPD: No